CLINICAL TRIAL: NCT00874172
Title: New Analgesic Strategy Combining Nitrous Oxide, Nefopam, Acetaminophen and Morphine Compared to the Usal Antalgic Strategy (Acetaminophen and Morphine) for the Treatment of Acute Sickle Cell Disease Pain in the Emergency Room
Brief Title: Effectiveness of New Analgesic Strategy Compared to the Usal Antalgic Strategy
Acronym: DREPANOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070605-OST07010
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-11

CONDITIONS: Sickle Cell Anemia
Keywords: Anemia; Sickle Cell; Analgesic; Pain; Emergency treatment; Quality of life
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Combination of acetaminophen, morphine
  Interventions: Drug: current analgesic strategy
- 1 (Experimental): Combination of acetaminophen, nitrous oxide, nefopam, morphine
  Interventions: Drug: Rapid optimized analgesic strategy

INTERVENTIONS:
Drug: Rapid optimized analgesic strategy — Oral treatment :
  1 gr Acetaminophen 20 mg of nefopam delivered on a lump sugar Nitrous oxide inhalation with initial output of 9 L/min subsequently Intravenous morphine bolus of 3 mg Nitrous oxide interruption after 5 minutes of the initial morphine bolus
  Arms: 1
Drug: current analgesic strategy — paracetamol 1 g per os nasal oxygen therapy
  1 amp of morphine 10 mg / 10 cc of glucose 5 %, by repeated bolus administration
  Arms: 2

SUMMARY:
Quality of life of adult patients with sickle cell disease is deeply impaired by severe adverse medical events that inadvertently occur throughout their time life. Indeed, patients not presenting a life threatening condition often present to the emergency department with sickle cell disease crisis related pain. Currently, the effectiveness of specific analgesic strategies for treating sickle cell disease crisis related pain are mostly based on acetaminophen and opioid derivates combination along with oxygen delivery. Those strategies are effective but may last up to half an hour to obtain pain relief. This delay mostly depends on the availability of venous access and on individual patient response to treatment. Nitrous oxide is a volatile efficient analgesic therapy that has been repeatedly shown to allow rapid analgesia in the emergency department setting.

The investigators hypothesise that a new analgesic strategy (rapid optimized analgesic strategy) including nitrous oxide and nefopam would be as safe and more rapidly effective than current analgesic strategy.

DETAILED DESCRIPTION:
Purpose of the study:

The main objective is to evaluate the effectiveness of an optimized combination of analgesic therapies for treating uncomplicated sickle cell disease crisis at initial visit to the emergency room of the Henri Mondor hospital.

Secondary objectives:

* Total amount of morphine required during the first 4 hours in the hospital emergency.
* Overall amount of morphine administered on the duration of patient stay in hospital Henri Mondor.
* Side effects of analgesic strategies
* Adverse medical events
* Length of hospital stay.
* 7-day and 1-month follow-up and collection of following data:

  1. Total number of sickle cell disease crises
  2. Number of subsequent readmission and/or visit to an ED
  3. Quality of life (EuroQol EQ-5D, and SF-36)
  4. Patient satisfaction: pain treatment satisfaction scale. Study design: prospective monocentric open-label randomized controlled trial Number of patients: 200 Follow up per patient: 1 month, Study enrolment period: 25 months.

Contraindications to nefopam administration: hypersensitivity to nefopam, benign prostatic hypertrophy and glaucoma, or history of seizures.

* contraindication to morphine administration hypersensitivity to morphine, decompensate respiratory failure, acute head trauma, uncontrolled epilepsy, severe hepatocellular failure, intracranial hypertension, use of buprenorphine or nalbuphine Contraindications to MEOPA administration, intra-cranial hypertension, non cooperative patient (sleepiness; encephalopathy, refusal to participate), pneumothorax, emphysema, pneumoperitoneum, digestive occlusion, pneumomediastinum, air embolism, diving accident , facial trauma, patients who recent administration of an ophthalmic gas (SF6, C3F8, C2F6) < 3 months).
* contraindication to the use of oxygen: no-absolute contraindication no health insurance, adults under tutelage

Main criterion:

Proportion of patients relieved (pain intensity by simple numerical scale <4) to 30 minutes of their arrival in the emergency department.

Secondary criteria:

* amount of morphine administrated within the first 4 hours of presentation to the emergency department
* overall amount of morphine administrated during hospital stay
* adverse event related with study treatment
* adverse medical events during hospitalization
* length of stay.
* 7-day and 1-month follow-up to collect the following data:

  1. Total number of sickle cell disease crises
  2. Number of subsequent readmission and/or visit to an ED
  3. Quality of life (EuroQol EQ-5D, and SF-36)
  4. Patient satisfaction: pain treatment satisfaction scale.

ELIGIBILITY:
Inclusion Criteria:

* male adult patient with sickle cell anemia,
* age ≥ 18 years,
* main complaint : sickle cell crisis pain,
* initial numeric pain intensity scale at presentation > 4,
* admission to the ED during working hours (amendment n°2-15/02/2010:from 8h to 20h), from Monday to Friday

Exclusion Criteria:

* female adult patient
* complicated sickle cell crisis or admission requirement to an ICU
* recent hospitalisation (< 10 days) for the same complaint
* previous inclusion in the study
* contraindication to anyone of the study drugs
* no medical insurance
* incompetent adult

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of pain relief (Numeric Pain Intensity Scale < 4) | at 30 min after admission to the ED

SECONDARY OUTCOMES:
Overall amount of morphine delivered | during the first 4 hours of ED presentation
Overall amount of morphine delivered | during the hospital stay following ED presentation and enrolment in the study
Analgesic drugs related adverse events | during the hospital stay following ED presentation and enrolment in the study
Length of hospital stay | during the hospital stay
Overall number of sickle cell crisis and patients'quality of life (EuroQol-EQ 5D, SF-36) and patients' satisfaction regarding pain management (pain management satisfaction questionnaire) | at 7 days and 30 days of follow-up.
measurement of oxygen saturation in tissue (amendment n°1 - 14/09/2009) | in 4hours after admission to the emergency
  measurement of oxygen saturation in tissue

CONTACTS AND LOCATIONS:
Overall Officials: Aline SANTIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Emergency Department, Créteil, France